CLINICAL TRIAL: NCT01440985
Title: An Evaluator-Blinded, Randomized, Parallel Controlled Study of Nicorette® Freshmint Gum Versus Nicorette® Microtab in Healthy Smokers Motivated to Quit Smoking With Visible Staining of Teeth
Brief Title: A Study on the Effects of Two Nicotine Replacement Products on Tooth Staining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: A6431085; 2005-001040-23 (EudraCT Number)
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Tooth Staining
MeSH Terms: conditions — Tobacco Use Disorder; Tooth Discoloration | interventions — Nicotine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine Gum (Experimental): After being randomized to the gum or tablet, dosage will be based on baseline level of nicotine dependence. Highly dependent smokers will receive nicotine 4 mg gum, while low nicotine-dependent smokers will receive nicotine 2 mg gum to help them quit. Subjects will be advised to use the treatment frequently, according to the product labeling, in order to minimize or avoid symptoms of tobacco withdrawal. Study medication will be used for 12 weeks.
  Interventions: Drug: Nicotine
- Nicotine Microtab (Active Comparator): After being randomized to the gum or tablet, subjects will receive instructions according to their baseline level of nicotine dependence. Highly dependent smokers will be instructed to use a 4 mg dosage of the Microtab (2 x 2 mg tablets), while low nicotine-dependent smokers will be instructed to use a 2 mg dosage of the Microtab to help them quit. Subjects will be advised to use the treatment frequently, according to the product labeling, in order to minimize or avoid symptoms of tobacco withdrawal. Study medication will be used for 12 weeks.
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Nicotine Gum 2 mg, Lot number GD922A
  Other Names: Nicorette® Freshmint Gum
  Arms: Nicotine Gum
Drug: Nicotine — Nicotine gum 4 mg, Lot number GC962A
  Other Names: Nicorette® Freshmint Gum
  Arms: Nicotine Gum
Drug: Nicotine — Nicotine Microtab 2 mg, Lot number GB196G
  Other Names: Nicorette® Microtab
  Arms: Nicotine Microtab

SUMMARY:
Participants will be smokers who want to quit, and have visible nicotine stains on their teeth. They will be given toothpaste and a toothbrush to use during the study, and will have an equal chance of being assigned to use either a nicotine gum or microtab. They will visit the study site five times during the 12 week trial to have their teeth examined.

DETAILED DESCRIPTION:
This evaluator-blinded, randomized, 12-week parallel-group controlled trial compares Nicorette® Freshmint gum versus Nicorette® Microtab in healthy smokers who are motivated to quit smoking and who have visible staining of teeth.

The trial is comprised of five visits (baseline, Weeks 1, 2, 6, and 12). At baseline, subjects will be provided with a standardized toothpaste and toothbrush; use of any other oral hygiene or tooth-whitening product is prohibited. At all visits after baseline, smoking status and use of study treatment will be checked. Teeth staining and teeth shade will be rated at baseline and at 2, 6 and 12 Weeks using the Modified Lobene Stain Index and the Vita® Shade Guide, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 65 years
* Daily smoker, current daily smoking for at least 1 year
* Motivated to quit smoking, and willing to use NRT (nicotine gum or nicotine sublingual tablet)
* Normal chewing abilities (able to use chewing gum without any problems)
* Willing to refrain from dental prophylaxis for the duration of the 12-week trial
* Have a minimum of 20 natural teeth, with at least 10 of the 12 anterior teeth present and scorable.
* Have a total extrinsic facial tooth stain score equal or more than 28, according to the MacPherson Modification of the Lobene Stain Index.
* Willing and able to comply with scheduled visits, treatment plan, tests, and other trial procedures.

Exclusion Criteria:

* Use of other tobacco-containing products, such as cigars, pipe, smokeless tobacco products, etc.
* Existing use of any nicotine replacement products for smoking cessation, or undergoing any other treatment for tobacco dependence, such as hypnosis, acupuncture, bupropion, etc.
* Orthodontic appliances
* Gross periodontal disease, or signs of gross oral neglect
* History of oral cancer
* History of temporomandibular joint disorders known to aggravate jaw pain
* Unstable angina pectoris or myocardial infarction during the previous 3 months
* Pregnancy, lactation or intended pregnancy
* Any major metabolic disease, clinically important renal or hepatic disease Suspected alcohol or drug abuse
* Participation in another clinical trial within the previous three months and during study participation
* Any other severe acute or chronic medical or psychiatric condition that might increase the risk associated with trial participation or trial drug administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, makes the subject inappropriate for entry into this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Total Extrinsic Tooth Stain Score | Baseline, 6 Weeks
  Mean change in total extrinsic tooth stain score, for the whole mouth region. Extrinsic tooth staining is measured using the MacPherson Modification of the Lobene Stain Index. A lower stain index score represents a reduction in extrinsic tooth staining.

SECONDARY OUTCOMES:
Change from Baseline in Total Extrinsic Tooth Stain Score | Baseline, 2 Weeks
  Mean change in total extrinsic tooth stain score, for the whole mouth region, measured using the MacPherson Modification of the Lobene Stain Index. A lower stain index score represents a reduction in extrinsic tooth staining.
Change from Baseline in Total Extrinsic Tooth Stain Score | Baseline, 12 Weeks
  Mean change in total extrinsic tooth stain score, for the whole mouth region, measured using the MacPherson Modification of the Lobene Stain Index. A lower stain index score represents a reduction in extrinsic tooth staining.
Change from Baseline in Mean Stain Index Facial Region | Baseline through Week 12
  Mean changes in the extrinsic facial surface stain score between baseline and Weeks 2, 6 and 12.
Change from Baseline in Mean Stain Index Lingual Region | Baseline through Week 12
  Mean changes in the extrinsic lingual surface stain score between baseline and 2, 6 and 12 weeks.
Change from Baseline in Mean Stain Index Body Region | Baseline through Week 12
  Mean changes in the extrinsic body region stain scores between baseline and 2, 6 and 12 weeks.
Change from Baseline in Mean Stain Index Gingival Region | Baseline through Week 12
  Mean changes in the extrinsic gingival region stain scores between baseline and 2, 6 and 12 weeks.
Change from Baseline in Mean Stain Index Interproximal Region | Baseline through Week 12
  Mean changes in the extrinsic interproximal region stain scores between baseline and 2, 6 and 12 weeks.
Change from Baseline in Mean Stain Area Total Region | Baseline through Week 12
  Mean stain area between baseline and Weeks 2, 6 and 12 for the facial region, lingual region, body region, gingival region, and interproximal region (Total Region).
Change from Baseline in Mean Stain Area Facial Region | Baseline through Week 12
  Mean stain area between baseline and Weeks 2, 6 and 12 for the facial region.
Change from Baseline in Mean Stain Area Lingual Region | Baseline through Week 12
  Mean stain area between baseline and Weeks 2, 6 and 12 for the lingual region.
Change from Baseline in Mean Stain Area Body Region | Baseline through Week 12
  Mean stain area between baseline and Weeks 2, 6 and 12 for the body region.
Change from Baseline in Mean Stain Area Gingival Region | Baseline through Week 12
  Mean stain area between baseline and Weeks 2, 6 and 12 for the gingival region.
Change from Baseline in Mean Stain Area Interproximal Region | Baseline through Week 12
  Mean stain area between baseline and Weeks 2, 6 and 12 for the interproximal region.
Change from Baseline in Mean Stain Intensity Total Region | Baseline through Week 12
  Mean stain intensity between baseline and Weeks 2, 6 and 12 for the facial region, lingual region, body region, gingival region, and interproximal region (Total Region).
Change from Baseline in Mean Stain Intensity Facial Region | Baseline through Week 12
  Mean stain intensity between baseline and Weeks 2, 6 and 12 for the facial region.
Change from Baseline in Mean Stain Intensity Lingual Region | Baseline through Week 12
  Mean stain intensity between baseline and Weeks 2, 6 and 12 for the lingual region.
Change from Baseline in Mean Stain Intensity Body Region | Baseline through Week 12
  Mean stain intensity between baseline and Weeks 2, 6 and 12 for the body region.
Change from Baseline in Mean Stain Intensity Gingival Region | Baseline through Week 12
  Mean stain intensity between baseline and Weeks 2, 6 and 12 for the gingival region.
Change from Baseline in Mean Stain Intensity Interproximal Region | Baseline through Week 12
  Mean stain intensity between baseline and Weeks 2, 6 and 12 for the interproximal region.
Change from Baseline in Mean Tooth Shade | Baseline through Week 12
  Mean tooth shade between baseline and Weeks 2, 6, and 12 using the Vita® Shade Guide. A higher number represents a lighter tooth shade.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- Dental School and Hospital, University College of Cork, Wilton, Cork, Ireland

REFERENCES:
- [Derived] Whelton H, Kingston R, O'Mullane D, Nilsson F. Randomized controlled trial to evaluate tooth stain reduction with nicotine replacement gum during a smoking cessation program. BMC Oral Health. 2012 Jun 13;12:13. doi: 10.1186/1472-6831-12-13. PMID 22695211